CLINICAL TRIAL: NCT00005345
Title: Genetic Epidemiology of Blood Lipids and Obesity - Ancillary to NGHS
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4212; R01HL045778 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Obesity

SUMMARY:
To conduct a genetic epidemiologic study of the coronary heart disease (CHD) risk factors of blood lipids and obesity in Black and white girls who participated in the NHLBI-supported National Growth and Health Study (NGHS). The study was ancillary to NGHS.

DETAILED DESCRIPTION:
BACKGROUND:

The National Growth and Health Study, NGHS, was an epidemiologic study of 2,379 black and white girls, ages 9-10 years at entry, who were followed annually. The ancillary study had the potential for identifying those genes involved in determining Black/white differences in lipid metabolism and obesity. This was an exciting area in which there was virtually no available information. Finally, the study permitted an examination of the effects of gene variation on changes in quantitative levels of blood lipids as well as in body fat during different stages of pubescence since the NGHS protocol included annual anthropometric and maturation assessments and biannual blood lipid determinations along with extensive environmental measures which included dietary, household, and psychosocial information. The study was unique because of the rare opportunity to do genetic analyses in a large cohort of two ethnic groups of children on whom a very rich data base was available.

DESIGN NARRATIVE:

The study was an independent research project ancillary to the NGHS and utilized the extensive biological and environmental information available from the NGHS core data base. Blood samples were obtained from 1,133 girls seen at their followup examinations in Year 7 in order to determine genotypes at those loci known to be implicated in lipid metabolism and obesity. Both protein [apolipoproteins C-II, D, and E and LP(a)] and DNA [apolipoprotein B, lipoprotein lipase (LPL), and LDL receptor] were analyzed. The distribution of genetic variation within each ethnic group was determined. At each candidate gene locus, the genotype effects were estimated on quantitative level of apolipoproteins and lipoproteins, and also on the degree and distribution of body fat after adjusting for concomitant variables (such as age, biologic maturation stage adiposity) within each ethnic group. By comparing the frequencies of genotypes at candidate loci, their allelic effects were assessed as well as their impact on blood lipids and obesity development in Black and white females.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-01; Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Kimm — University of Pittsburgh

REFERENCES:
- [Background] Kimm SY, Pasagian-Macaulay A, Aston CE, McAllister AE, Glynn NW, Kamboh MI, Ferrell RE. Correlates of lipoprotein(a) levels in a biracial cohort of young girls: the NHLBI Growth and Health Study. J Pediatr. 1999 Aug;135(2 Pt 1):169-76. doi: 10.1016/s0022-3476(99)70018-1. PMID 10431110
- [Background] Sanghera DK, Ferrell RE, Aston CE, McAllister AE, Kamboh MI, Kimm SY. Quantitative effects of the apolipoprotein E polymorphism in a biracial sample of 9-10-year-old girls. Atherosclerosis. 1996 Sep 27;126(1):35-42. doi: 10.1016/0021-9150(96)05891-1. PMID 8879432
- [Background] Hagberg JM, Moore GE, Ferrell RE. Specific genetic markers of endurance performance and VO2max. Exerc Sport Sci Rev. 2001;29(1):15-9. doi: 10.1097/00003677-200101000-00004. PMID 11210441
- [Background] Moffett S, Martinson J, Shriver MD, Deka R, McGarvey ST, Barrantes R, Ferrell RE. Genetic diversity and evolution of the human leptin locus tetranucleotide repeat. Hum Genet. 2002 May;110(5):412-7. doi: 10.1007/s00439-002-0715-5. Epub 2002 Apr 4. PMID 12073010